CLINICAL TRIAL: NCT00002880
Title: PHASE II STUDY OF ORAL ETOPOSIDE WITH PHARMACODYNAMIC MODELING IN RELAPSED NON-HODGKIN'S LYMPHOMA (IWF GRADES A-H)
Brief Title: Etoposide in Treating Patients With Relapsed Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-9650; U10CA031946 (NIH); CLB-9650; CDR0000065180 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Lymphoma
Keywords: Waldenstrom macroglobulinemia; recurrent small lymphocytic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic | interventions — etoposide phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etoposide (Experimental): Oral etoposide for relapsed or refractory non-Hodgkin's lymphoma
  Interventions: Drug: Etoposide phosphate

INTERVENTIONS:
Drug: Etoposide phosphate — 50 mg PO q day for 21 days; repeat every 28 days escalate dose to 100 mg PO q day if ANC remains greater than 1500/microliter during cycle 1: no specified maximum of cycles if PR or CR

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of etoposide in treating patients with relapsed non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the response rate and response duration in patients with relapsed non-Hodgkin's lymphoma when treated with daily oral etoposide. II. Describe the toxic effects of daily oral etoposide in these patients. III. Monitor etoposide trough levels and determine whether etoposide concentrations correlate with age, response, and toxicity.

OUTLINE: Patients receive oral etoposide daily for 21 days. Treatment is repeated every 28 days in the absence of disease progression or unacceptable toxicity. Patients in complete or partial remission receive 2 courses past best response (minimum 6 courses). Patients with stable disease after 3 courses may be removed from study. Patients are followed every 6 months for 2 years, then annually for survival.

PROJECTED ACCRUAL: Approximately 97 patients will be accrued for this study over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically documented non-Hodgkin's lymphoma Needle or core biopsy not acceptable as sole means of diagnosis No mantle cell or transformed lymphoma One of the following International Working Formulation (IWF) histologic subtypes required: Small lymphocytic with absolute lymphocytic count less than 5,000 (IWF A) Follicular, predominately small cleaved cell (IWF B) Follicular, mixed (IWF C) Follicular, large cell (IWF D) Diffuse, small cleaved cell (IWF E) Diffuse, mixed (IWF F) Diffuse, large cell (IWF G) Large cell, immunoblastic (IWF H) Recurrent or refractory disease treated with no more than 4 prior chemotherapy regimens Rebiopsy of a node at first relapse recommended Prior etoposide (oral or intravenous) allowed if given for no more than 5 days every 3 weeks The following are considered 1 prior therapy each: Identical drugs given on 2 different schedules Bone marrow transplant preparative regimen (single cycle of chemotherapy used solely to mobilize peripheral blood stem cells considered part of preparative regimen) Ineligible for protocol CLB-9551 (aminocamptothecin) Measurable disease by physical exam or imaging study required Indicator lesion larger than 1 x 1 cm No prior radiotherapy to indicator lesion unless progression clearly documented The following are not considered measurable: Barium study Ascites or pleural effusions Bony disease Bone marrow involvement No known parenchymal or leptomeningeal CNS disease Lumbar puncture not required prior to study

PATIENT CHARACTERISTICS: Age: Not specified Performance status: CALGB 0-2 Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times normal Renal: Creatinine no greater than 1.5 times normal Other: HIV negative (testing required for patients at risk) No uncontrolled infection No other serious medical condition that would interfere with evaluation of study agent No psychiatric condition that would preclude protocol completion or informed consent No second malignancy within 5 years except curatively treated: Basal cell skin cancer Cervical cancer Not pregnant or nursing Adequate contraception required of fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 3 weeks since prior chemotherapy (3 weeks for nitrosoureas, melphalan, or mitomycin) Endocrine therapy: No concurrent corticosteroids except for physiologic replacement Radiotherapy: At least 3 weeks since prior radiotherapy Surgery: Not specified Other: No other concurrent investigational agent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 1996-11; Primary Completion 2001-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics of etoposide | days 8, 15, and 22 of tx

SECONDARY OUTCOMES:
Response | Day 1 of ea cycle, then q 6 mon/2 yrs then yearly until death or ds progression

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Bartlett, MD, Study Chair — Washington University Siteman Cancer Center
Locations (4):
- United States (4):
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Washington University Barnard Cancer Center, St Louis, Missouri
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina